CLINICAL TRIAL: NCT05506059
Title: "BES2T" (Bedside E-point Septal Separation Test) for Emergency Medicine Residents
Brief Title: Heart Ultrasound by Emergency Medicine Residents as an Estimate of Heart Function
Acronym: BES2T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Guthrie Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2206-26
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Stroke Volume; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The doctor's doing the ultrasounds will be blinded to each other's measurements and to the patient's past medical history
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Volunteer (Other): Healthy volunteers over the age of 18 who consent to two ultrasounds.
  Interventions: Diagnostic Test: Ultrasound
- ED patient with planned heart echocardiogram (Experimental): Patients in emergency department (ED) who have a heart echocardiogram scheduled as part of their routine clinical care
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Participants will have ultrasounds of the heart by two different emergency medicine doctors.

SUMMARY:
The purpose of this research is to better understand the use of heart ultrasounds to estimate heart function.

DETAILED DESCRIPTION:
This research involves ultrasounds of the heart by two different emergency medicine doctors who are residents in training. Results from the two doctors will be compared to see how similar they are. This research will help us understand if heart ultrasounds can be used to see how well the heart pumps blood and if similar results are obtained from different doctors.

The doctors will use ultrasound of the heart to measure E-Point Septal Separation (EPSS). EPSS is the distance between two parts of the heart, the mitral valve and the ventricular septum. EPSS is measured in millimeters (mm). EPSS can estimate left ventricular ejection fraction (LVEF) as a measure of how well the heart pumps blood.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, or patients who come to the emergency department who may have a heart echocardiogram scheduled as part of their routine clinical care
* Age 18 or over
* Willing and able to provide informed consent

Exclusion Criteria:

* Pediatrics (age <18 years old).
* No cardiac-altering intervention performed between examiners.
* Unable to obtain a parasternal long view with mitral valve anterior leaflet, interventricular septum and aortic root.
* Transthoracic echocardiogram (TTE) more than the next day after EPSS is performed (for secondary outcome).
* Female with known pregnancy.
* Prisoner
* Prior cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-09-10 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Mean change in millimeters between E-Point Septal Separation (EPSS) measurements of the heart by two physicians | During procedure
  Two physicians will use the same ultrasound device to measure the E-Point Septal Separation (EPSS) on the same patients. EPSS is the distance between two parts of the heart, the mitral valve and the ventricular septum. The mean change in EPSS measurements in millimeter will be calculated.

SECONDARY OUTCOMES:
Percent change in Left Ventricular Ejection Fraction (LVEF) estimated from ultrasound compared to a formal transthoracic echocardiogram. | During procedure
  Percent change in Left Ventricular Ejection Fraction (LVEF) estimated from ultrasound compared to a formal transthoracic echocardiogram. LVEF (in %) will be estimated from ultrasound using the formula = 75.5 - (2.5 x E-Point Septal Separation in millimeters)

CONTACTS AND LOCATIONS:
Overall Officials: Dean Licurgo, DO, Principal Investigator — The Guthrie Clinic
Locations (1):
- The Robert Packer Hospital, Sayre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No